CLINICAL TRIAL: NCT03108859
Title: Pre-and In-hospital First Aid Programs and Specifications for Spine and Spinal Cord Injury in Beijing of China: a Prospective, Multicenter, Case Series Trial
Brief Title: Pre-and In-hospital First Aid Programs and Specifications for Spine and Spinal Cord Injury in Beijing of China
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Baoguo Jiang, Principal Investigator, Peking University People's Hospital
Other Study IDs: PekingUPH_002
Record Dates: First submitted 2017-04-06; First posted 2017-04-11 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To establish a spine injury and spinal cord injury (SCI) treatment database; to complete pre- and in-hospital evaluation of spine injury and SCI, develop and optimize first aid procedures, form pre-and in-hospital standardized training program for the treatment of spine injury and SCI; to develop first aid guidelines and establish an evaluation and treatment system for early surgery, as far as possible to save the spinal cord function and reduce the degree of disability; to form expert consensus on acute SCI and "green channel" patterns, will be promoted in hospitals in Beijing and other cities of China, so as to improve the level of first aid treatment of acute spine injury and SCI in Chinese cities, and to reduce the occurrence of secondary injury and severe dysfunction due to improper treatment.

DETAILED DESCRIPTION:
This is a prospective, multicenter, non-randomized controlled trial. The target population consists of 200 acute spinal cord injury patients undergoing pre-hospital treatment in the Beijing Emergency Medical Center and Beijing Red Cross Emergency Rescue Center, and receiving in-hospital treatment in the Peking University People's Hospital, Peking University Third Hospital, Beijing Friendship Hospital Affiliated to Capital Medical University, Chaoyang Hospital Affiliated to Capital Medical University, and Chinese PLA General Hospital, China.

History and current related studies Acute spinal cord injury (SCI) as a clinical common disease is the difficulty of clinical treatment, and frequently occurs in young adults. The incidence of acute SCI is 30-40/million people in Europe and USA, but 60.2/million people in Beijing of China. The complete SCI is very dangerous, and there is no effective medical therapy. At present, the effective treatment of acute SCI should be the first aid and advanced rehabilitation.

24 hours is the best time to rescue spinal cord function after SCI, especially 3-8 hours after injury is the golden opportunity. A large dose of hormone therapy in the 3-8 hours after injury can reduce secondary injury, thereby reducing the degree of SCI. 24 hours after injury, early surgery for relieving spinal cord compression can significantly improve the recovery of spinal cord function. Timely and properly pre-hospital first aid, quick hospital admissions and assessment, and timely surgery are essential for the rescue of spinal cord function. Patients with incomplete SCI can be completely injured and lose the possibility of recovery of spinal cord function due to improper first aid or untimely treatment. Complete SCI will cause more severe injury due to improper treatment. It may be difficult to make up for surgery or rehabilitation training. A sound and rapid treatment system is the basis for improving the treatment level of SCI, but we still lack of this kind of system in China.

In Beijing of China, pre-hospital treatment can be done by Beijing Emergency Medical Center (120 first aid system) and Beijing Red Cross Hospital (999 first aid system). While cooperating with each other, it is also faced with different mechanisms, different treatment patterns and overlapping treatment regions. As for the in-hospital treatment, Beijing has a large number of high-level hospitals, but these hospitals are overcrowding. There is no SCI treatment specialist or professional hospital in Beijing City, so treatment basically relies on various general hospitals. In pre-hospital first aid and in-hospital treatment of Beijing City, the medical information transfer is not smooth; the treatment process is separated, and it lacks of standardized treatment. The ability and level of medical personnels are not consistent, the technology is backward, and there is lack of professional training. Thus, the vast majority of patients with SCI cannot be treated within the optimal treatment time after injury. It is also an important cause of higher mortality and disability in SCI patients in China compared with the developed countries.

In 2006, Professor Bao-guo Jiang, director of the Department of Orthopedics, Peking University People's Hospital, led the establishment of the Traffic Medicine Center of Peking University, involving Peking University People's Hospital, School of Public Health of Peking University, Peking University First Hospital, Peking University Third Hospital, Beijing Traffic Management Bureau, and Beijing Emergency Medical Center in China. Reviewed by the Health and Family Planning Commission, the "National Center for Severe Trauma Training" was set up in 2015, and Bao-guo Jiang served as the director of the center. The Traffic Medicine Center and two emergency centers in Beijing have cooperated for many years, and established an epidemiological database for the treatment of severe trauma and the linkage mechanism of pre-hospital and in-hospital. The treatment of spine injury and SCI is one of important contents for treating severe trauma. With this center as a platform, the database of SCI patients can be specialized; a unified standardized and rapid treatment can be carried out in many participating medical units using the linkage mechanism with the emergency centers; a high level of scientific research can be carried out, and a series of studies can be started, concerning SCI epidemiology, treatment procedures and improvement in treatment effect. Simultaneously, the standardized training for pre-hospital and in-hospital first aid care personnel in each research center and hospital can be completed.

For nonstandard treatment process and path and poor information exchange, incoherent pre-hospital care and in-hospital treatment, lack of professional training for treatment personnel, and uneven comprehensive hospital treatment capacity, this trial aims to formulate the standards for the treatment of spine injury and SCI through a standardized multicenter study so as to improve the level of SCI treatment and to reduce the mortality and disability of SCI patients in Beijing, China.

Statistical analysis

1. Statistical analysis will be performed using SPSS 19.0 software (IBM, Armonk, NY, USA)
2. Measurement data will be expressed as the case number (missing number), mean, median, standard deviation, first quartile, third quartile, maximum, and minimum. The 95% confidence interval of the rate will be calculated.
3. Count data will be expressed as the frequency and relative number. The 95% confidence interval of the rate will be calculated.
4. Normally or non-normally distributed measurement data will be analyzed using paired t-test or Wilcoxon signed rank test.
5. Count data will be analyzed using Chi-square test or Fisher exact test. Ranked data will be analyzed using Wilcoxon signed rank test.

Sample size calculation In accordance with previous SCI treatment conditions in participating units, we will recruit 200 cases.

Data management

1. The database will be constructed and maintained by Peking University People's Hospital. According to the data characteristics of the research program, the main researcher will draft detailed data management and statistical plans, including data quality audit, construct corresponding electronic database, completely and accurately input all expected data.
2. Each participating unit will be responsible for filling in the database of their subjects.
3. The computer program combined with the manual method will be used to check the consistency and logicality of the data.
4. Any questions will be answered by the person in charge of the project and the main staff, and returned to the data management center, and then the data manager will modify and update the database. All inspection procedures need to be repeated several times until there is no doubt. All changes and updates are required for recording and filing. It is strictly forbidden to use correction fluid or correction tape.
5. All researchers are required to ensure that the data recorded in the case report forms are authentic.

Auditing

1. Peking University People's Hospital will organize training sessions before the study and conduct unified training for all the participants. A person, as a coordinator, will coordinate the whole research, prepare a research brief, regularly announce the progress of the study, and solve the problems in the study.
2. The responsible person will hold a regular meeting, summarize the work, communicate, correct the problem, and make a request.
3. In order to follow the Guidelines for Good Clinical Practice, we will set up a regular visit to each center to ensure compliance with research programs, Good Clinical Practice and related laws.

Quality control and management

1. In order to implement the research plan, it is necessary to hold the project launch meeting of the heads of the participating units so as to carry out unified training for the implementation of the project plan, and for the record and assessment.
2. The heads of the participating units will train specific operators on programs, procedures, and instructions, develop training programs and manuals to ensure that the team members are familiar with and grasp the relevant contents before the trial.
3. The inspector is responsible for ensuring the smooth progress of the trial, controls the whole process, and deals with emergencies.
4. Each participating unit will perform its duties, strictly follow the clinical trial program, and adopt standard operating procedures. Grading of quality-control staffs will be set up; different grades of staffs will be responsible for different parts of work, which will be inspected by the superior staff to ensure that the data will be input in the database system within 24 hours after the incident and to ensure the authenticity and validity.
5. A new team member will be trained, concerning project plan and process, and timely trained, concerning the updated content/process or content that needs to be re-emphasized.
6. Standard operation procedure will ensure smooth handover if necessary.
7. The arbitrator will guarantee the rights of each participating unit, make sure true, accurate, complete and correct data record and report, and ensure that the research follows the relevant laws and regulations. The number of visits of the arbitrator will meet the needs of quality control. The arbitrator after each visit will inform the project leader the inspection results.
8. Quality controller of each region will carry out internal inspection on scale filling weekly according to the requirements.
9. According to the training program, the leader of each region will submit the results, statements, and a summary report quarterly to the research group. The research group will timely adjust the protocol according to the report.

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord injury patients will be evaluated as complete or incomplete (contusion) after admission using rectal examination, in accordance with American Spinal Injury Association and International Medical Society of Paraplegia (2000);
* Final diagnosis by spine CT and/or MRI;
* Cervical, thoracic and thoracolumbar fracture dislocation or without fracture dislocation but combined with spinal cord injury;
* No other injury involving life, injury severity score < 16;
* No anesthesia contraindication;
* No local skin infection, no severe soft tissue contusion, soft tissue condition of the operation area met the operation requirements;
* Age: 16-85 years old, irrespective of sex.

Exclusion Criteria:

* Active or recent severe infection
* Severe infectious diseases that need to be treated in infectious disease hospital;
* History of mental illness;
* History of metal allergy;
* Long-term alcohol abuse and drug abuse;
* Do not agree to participate in this trial; the legal representative of the patient refuses to sign informed consent;
* Poor compliance, cannot be followed up as required.

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: To recruit acute SCI patients undergoing pre-hospital treatment in the Beijing Emergency Medical Center and Beijing Red Cross Emergency Rescue Center, and receiving in-hospital treatment in the Peking University People's Hospital, Peking University Third Hospital, Beijing Friendship Hospital Affiliated to Capital Medical University, Chaoyang Hospital Affiliated to Capital Medical University, and Chinese PLA General Hospital, China.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-05 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
American Spinal Injury Association impairment scale | changes of week 1, month 1 and month 3 after surgery
  To assess spinal nerve function at postoperative 1 week, 1 and 3 months

SECONDARY OUTCOMES:
X-ray, spine CT and MRI scans | changes of week 1, month 1 and month 3 after surgery
  To assess spine injury and SCI and repair at preoperative, postoperative 1 week, 1 and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Baoguo Jiang, Ph.D, Principal Investigator — Department of Orthopedics, Peking University People's Hospital, Beijing, China
Locations (4):
- China (4):
  - Chaoyang Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality
  - Beijing Friendship Hospital Affiliated to the Capital University of Medical Sciences, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Undecided